CLINICAL TRIAL: NCT01972984
Title: The NEO (NEOADJUVANT ENDOCRINE OUTCOMES) TRIAL: Neoadjuvant Endocrine Therapy for Primary Breast Cancer: Investigation of Clinical and Translational Outcomes
Brief Title: Feasibility Study of Presurgical Hormone Therapy (Anastrozole) in Breast Cancer Patients
Acronym: NEO ER 11-05
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011712-01H
Record Dates: First submitted 2013-09-26; First posted 2013-10-31 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: Estrogen receptor positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anastrozole (Experimental): All qualifying women will receive anastrozole at the usual dose of 1mg daily for 2-6 weeks leading up to their surgery
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Anastrozole — Participants will be instructed to take one tablet of anastrozole orally per day with fluids. This tablet will be taken at the same time every day. Participants will be given a drug diary to record drug administration and aid in drug compliance. Should the participant miss a dose they will be asked to record it in their diary and resume the normal dose schedule the next day.
  Other Names: Arimidex

SUMMARY:
1. Women with operable breast cancer with a 2-8 week preoperative waiting period will accept preoperative therapy trials and specifically taking a standard drug for breast cancer such as anastrozole in this study
2. Short term anastrozole treatment will induce measurable changes in biomarker levels (ER, PR, Her2, Ki67) within the tumor.
3. Degree of response to short term anastrozole varies with a) duration of treatment and b) breast cancer subtype (based on initial pre-treatment biomarker status)

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed postmenopausal women (Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 20 pg/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago.)
2. Confirmation of estrogen receptor positive invasive carcinoma on core biopsy
3. Patients whose cancers are palpable and have been deemed to be "operable" by the surgeon
4. Surgery is planned for the next 2-8 weeks.

Exclusion Criteria:

1. History of hormone replacement therapy in the last 6 months
2. Previous treatment by tamoxifen or aromatase inhibitor treatment in six months
3. Known hypersensitivity or contraindications to aromatase inhibitors
4. Known metastatic disease on presentation
5. Recurrent breast cancer
6. Inability to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who fit the eligibility criteria that consent to the study; withdraw after consent from the study. | up to 18 months
  Participants are on study from the time their eligibility is confirmed until the time of their surgery which could be up to 8 weeks. This is a feasibility study and therefore once the study is closed to accrual the percent of women who signed consent and remained on study until their surgery versus those who withdraw will be determined.

SECONDARY OUTCOMES:
Measure the changes in ER, PR, Her2 and Ki67 labelling index on pre- and post treatment tumor tissue | Up to 18 months
  All biomarker results will be analyzed at study closure when participant #20 has received surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Arnaout, Dr., Principal Investigator — The Ottawa Hospital Cancer Centre
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada